CLINICAL TRIAL: NCT01159379
Title: Cross-reactivity and Tolerability of Ertapenem in Patients With IgE-mediated Allergy to Beta-lactams
Brief Title: Safety of Ertapenem in Beta-lactam Allergic Patients.
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Catholic University of the Sacred Heart (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Prof. Domenico Schiavino, Catholic University of the Sacred Heart
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 1131/09
Record Dates: First submitted 2010-06-03; First posted 2010-07-09 (Estimated); Last update posted 2011-01-05 (Estimated); Status verified 2010-01

CONDITIONS: IgE-Mediated Hypersensitivity; Allergy
Keywords: IgE-mediated allergy; Beta-lactams; Ertapenem; Cross-reactivity; Immediate-type skin tests; Intravenous tolerance tests
MeSH Terms: conditions — Hypersensitivity, Immediate; Hypersensitivity | interventions — Ertapenem

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- ertapenem, tolerance tests (Experimental): Patients with IgE-mediated allergy to beta-lactams
  Interventions: Drug: ertapenem

INTERVENTIONS:
Drug: ertapenem — intravenous, 1 gram, once
  Other Names: Invanz

SUMMARY:
The purpose of this study is to assess cross-reactivity and tolerability of ertapenem in patients with IgE-mediated allergy to at least one beta-lactam molecule.

DETAILED DESCRIPTION:
Ertapenem is a new carbapenem, stable to dehydropeptidase which has a broad antibacterial activity. Ertapenem exhibits a bactericidal mode of action and it has a long half-life of 4.5 hours; for this reason it can be developed as a single daily dose carbapenem.

In literature, no cases of IgE-mediated allergy to ertapenem have been described until now. However, a single study put in evidence a 47% rate of cross-reactivity between imipenem-cilastatin and beta-lactams in a group of patients affected by IgE-mediated allergy to these drugs. For this reason carbapenem administration to beta-lactam allergic patients has always been considered potentially harmful. Other studies reported lower cross-reactivity rates (from 7 to 11%) between imipenem-cilastatin and beta-lactams but patients of these studies did not undergo any allergy testing in order to demonstrate the pathogenesis of the reactions.

Recent studies put in evidence that imipenem has a very low cross-reactivity rate with other beta-lactams and they have a very good tolerability among patients with IgE-mediated allergy to beta-lactams: Romano et al. found a cross-reactivity rate of 0.9% between imipenem and penicillins in 112 penicillin-allergic patients (mean age 44.56 ± 15.66 ys.); Atanasković-Marković et al. found a cross-reactivity rate of 0.8% in 124 paediatric patients (age range 3-14 ys.) between imipenem and penicillins. In both groups imipenem was well tolerated by patients with negative allergy testing.

Meropenem showed to have a good tolerability too in penicillin allergic patients: Romano et al. found a cross-reactivity rate of 0.9% between penicillins and meropenem in penicillin-allergic patients (mean age 47.83 ± 15.8); Atanasković-Marković et al. found a cross-reactivity rate of 0.8% in 109 paediatric patients (age range 3-14 ys.) between meropenem and penicillins. In both groups meropenem was well tolerated by patients with negative allergy testing.

No data regarding the cross-reactivity of ertapenem with other beta-lactams and its tolerability among patients with IgE-mediated allergy beta-lactams are available in literature.

Aim of the study On the basis of those data, we decided to investigate the cross-reactivity of ertapenem with other beta-lactams in patients suffering from IgE-mediated allergy to at least one beta-lactam molecule and its tolerability in a group of a patients with negative allergy testing with ertapenem.

ELIGIBILITY:
Inclusion Criteria:

* IgE-mediated allergy to at least one beta-lactam molecule

Exclusion Criteria:

* positive allergy testing to ertapenem
* chronic diseases
* treatment with beta-blockers
* pregnancy

Ages: 16 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2011-01; Primary Completion 2011-09 (Estimated); Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
Cross-reactivity between beta-lactams and ertapenem. | 1 day

SECONDARY OUTCOMES:
Tolerability of ertapenem in patients with IgE-mediated allergy to beta-lactams. | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Domenico Schiavino, MD, Principal Investigator — Allergy Department, Catholic University of the Sacred Heart
Locations (1):
- Allergy Department, Catholic University of the Sacred Heart, Rome, Italy